CLINICAL TRIAL: NCT02731820
Title: Efficacy of Potassium Citrate in the Treatment of Postmenopausal Osteopenia. A Randomized, Placebo-controlled, Double Blind Investigation.
Brief Title: Efficacy of Potassium Citrate in the Treatment of Postmenopausal Osteopenia
Acronym: ACAROS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Principal Investigator, Nicola Baldini, MD, Professor, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 6013_IOR; 1676 (Other: Istituto Ortopedico Rizzoli)
Record Dates: First submitted 2016-03-31; First posted 2016-04-08 (Estimated); Results first posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-10

CONDITIONS: Osteopenia; Bone Disease, Metabolic
Keywords: potassium citrate
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — Potassium Citrate; Cholecalciferol; Calcium Carbonate

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Treatment group (Experimental): Potassium citrate Calcium carbonate Vitamin D3
  Interventions: Dietary Supplement: Potassium citrate; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate
- Control group, Placebo (Placebo Comparator): Placebo (Excipients) Calcium carbonate Vitamin D3
  Interventions: Dietary Supplement: Placebo; Dietary Supplement: Vitamin D3; Dietary Supplement: Calcium carbonate

INTERVENTIONS:
Dietary Supplement: Potassium citrate — Kcitr 3.064 milligrams daily in two tablets by mouth (1.032 milligrams every 12 hours)
  Arms: Treatment group
Dietary Supplement: Placebo — Excipients: 3.064 milligrams daily in two tablets by mouth (1.032 milligrams every 12 hours)
  Arms: Control group, Placebo
Dietary Supplement: Vitamin D3 — 400 IU/die Vitamin D3 daily by mouth
  Other Names: Cholecalciferol
Dietary Supplement: Calcium carbonate — 500 mg/die calcium carbonate daily by mouth

SUMMARY:
The purpose of this study is to investigate whether the use of alkali compounds, i.e. potassium citrate (K3C6H5O7, hereinafter KCitr) is effective in preventing the progression of osteopenia.

A randomized clinical trial (RCT, placebo-controlled, double-blind) has been planned to evaluate the effect of the daily administration of KCitr (3 g/die, K 30 mEq).

The efficacy will be evaluated by comparing the circulating levels of bone turnover markers at the baseline and after the treatment (3, 6 months).

DETAILED DESCRIPTION:
Bone tissue carries out some of the important metabolic functions, including the regulation of acid-base balance. In order to buffer the systemic acidosis, the skeleton acts as a "ion exchange column" modifying the composition of the mineral portion, i.e. the hydroxyapatite. There is a linear correlation between elimination of calcium and acidosis: the higher is the acidosis, the higher will be the loss of calcium from bones. In vitro experiments showed that acidosis also directly influences the cellular component of bone by increasing the osteoclast activity and inhibiting the production of the mineralized matrix by osteoblast. Since the low pH is a risk factor that accelerates the bone loss, the use of alkalizing compounds could prevent the osteopenia or support the conventional therapy of the osteoporosis.

KCitr is an alkaline compound which may be used in metabolic acidosis. Potassium is an alkaline metal that plays a pivotal role in the function of all living cells. Citric acid is a key molecule of the Krebs cycle, and it is abundant in bone where exhibits a stabilizing function. Although clinical data regarding the KCitr effectiveness on calcium metabolism are encouraging, it is still unclear whether the beneficial effects are due exclusively to the buffering function or whether KCitr may affect the bone cells activity. The purpose of this study is to evaluate the effects of KCitr on bone metabolism. We hypothesize that administration of potassium citrate to postmenopausal women with osteopenia will delay (or will prevent) the weakening of bone mass.

Postmenopausal women with osteopenia (T score between -1.0 and -2.5) and no history of fracture will be randomized to assume KCitr ate or placebo, daily for six months. Primary outcomes will be evaluated by measuring markers of bone turnover, which will be measured at baseline (before treatment), in the mid-term (3 months) and at the end (6 months).

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women, more than 5 years post menopause
* Osteopenia (T-score < -1 and > -2.5)
* Low risk of fracture (FRAX: < 20 major osteoporotic; < 3 hip fracture)

Exclusion Criteria:

* Hyperkalemia
* Renal insufficiency
* Nephrolithiasis
* Use of potassium sparing diuretics
* Use of potassium supplements
* Use of therapies influencing bone metabolism (e.g. corticosteroids, thiazide diuretics, aromatase inhibitors, estrogens)
* Use of protonic pump inhibitors
* Current or recent use of bisphosphonates (stopped less than three years prior to the start of the study)
* Gastrointestinal disorders that hamper nutrient absorption;
* Mental or psychiatric disorders that preclude the possibility of correctly adhering to the protocol

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2015-09-01 (Actual); Primary Completion 2017-08-30 (Actual); Study Completion 2017-09-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nicola Baldini, MD, Prof., Principal Investigator — Istituto Ortopedico Rizzoli
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Italy

IPD SHARING:
Plan to Share IPD: No
All the results will be available "on request"

REFERENCES:
- [Background] Arnett TR. Acidosis, hypoxia and bone. Arch Biochem Biophys. 2010 Nov 1;503(1):103-9. doi: 10.1016/j.abb.2010.07.021. Epub 2010 Jul 23. PMID 20655868
- [Background] Lambert H, Frassetto L, Moore JB, Torgerson D, Gannon R, Burckhardt P, Lanham-New S. The effect of supplementation with alkaline potassium salts on bone metabolism: a meta-analysis. Osteoporos Int. 2015 Apr;26(4):1311-8. doi: 10.1007/s00198-014-3006-9. Epub 2015 Jan 9. PMID 25572045
- [Background] Hanley DA, Whiting SJ. Does a high dietary acid content cause bone loss, and can bone loss be prevented with an alkaline diet? J Clin Densitom. 2013 Oct-Dec;16(4):420-5. doi: 10.1016/j.jocd.2013.08.014. Epub 2013 Oct 2. PMID 24094472
- [Background] Jehle S, Hulter HN, Krapf R. Effect of potassium citrate on bone density, microarchitecture, and fracture risk in healthy older adults without osteoporosis: a randomized controlled trial. J Clin Endocrinol Metab. 2013 Jan;98(1):207-17. doi: 10.1210/jc.2012-3099. Epub 2012 Nov 15. PMID 23162100
- [Result] Granchi D, Caudarella R, Ripamonti C, Spinnato P, Bazzocchi A, Massa A, Baldini N. Potassium Citrate Supplementation Decreases the Biochemical Markers of Bone Loss in a Group of Osteopenic Women: The Results of a Randomized, Double-Blind, Placebo-Controlled Pilot Study. Nutrients. 2018 Sep 12;10(9):1293. doi: 10.3390/nu10091293. PMID 30213095
- See also: Istituto Ortopedico Rizzoli_Home Page — http://www.ior.it/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited among the cohort of post-menopausal women attending to the Radiodiagnostic Unit of Istituto Ortopedico Rizzoli (IOR) from September 2015 to February 2017 to perform the periodic measurements of lumbar (at L2-L4 level) and femoral bone mineral density (BMD) by dual-energy X-ray absorptiometry (DXA).
Groups:
- Treatment Group, Potassium Citrate: Potassium citrate Calcium carbonate Vitamin D3
  Potassium citrate: Kcitr 3.064 milligrams daily in two tablets by mouth (1.032 milligrams every 12 hours)
  Vitamin D3: 400 IU/die Vitamin D3 daily by mouth
  Calcium carbonate: 500 mg/die calcium carbonate daily by mouth
Period: Overall Study
Arm/Group | Treatment Group, Potassium Citrate | Control Group, Placebo
Started | 20 | 20
Completed | 17 | 18
Not Completed | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Treatment Group, Potassium Citrate | Control Group, Placebo | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 60.8 (4.67) | 58.2 (4.95) | 59.5 (4.93)
Sex: Female, Male [Count of Participants; unit: Participants] — Osteopenic post-menopausal women
  Participants
    Female | 20 | 20 | 40
    Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 20 | 20 | 40
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 20 | 20 | 40
Region of Enrollment [Number; unit: participants]
  Italy | 20 | 20 | 40
Body mass index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 23.6 (4.4) | 22.9 (3.8) | 23.3 (4.1)
T score (BMD femural neck) [Mean (Standard Deviation); unit: scores on a scale] — T-score shows how much bone mineral density (BMD) is higher or lower than the bone density of a healthy 30-year old adult.
  According to the World Health Organization (WHO):
  * T-score of -1.0 or above= normal bone density;
  * T-score between -1.0 and -2.5 means = osteopenia;
  * T-score of -2.5 or below = osteoporosis.
  scores on a scale | -1.6 (0.4) | -1.7 (0.5) | -1.6 (0.5)
T score (L2 - L4) [Mean (Standard Deviation); unit: scores on a scale] — T-score shows how much bone mineral density (BMD) is higher or lower than the bone density of a healthy 30-year old adult.
  According to the World Health Organization (WHO):
  * T-score of -1.0 or above= normal bone density;
  * T-score between -1.0 and -2.5 means = osteopenia;
  * T-score of -2.5 or below = osteoporosis.
  scores on a scale | -1.7 (0.5) | -1.4 (0.6) | -1.6 (0.6)
Major osteoporotic risk [Mean (Standard Deviation); unit: % (percentage probability)] — Ten-year percentage probability of a major osteoporotic fracture (spine, forearm, hip or shoulder fracture) calculated according to "Fracture risk assessment tool (FRAX™)" (available on www.sheffield.ac.uk/FRAX/tool.aspx?lang=en).
  % (percentage probability) | 5.7 (3.4) | 4.8 (1.5) | 5.2 (2.6)
Minor osteoporotic risk [Mean (Standard Deviation); unit: % (percentage probability)] — Ten-year percentage probability of hip fracture calculated according to "Fracture risk assessment tool (FRAX™)" (available on www.sheffield.ac.uk/FRAX/tool.aspx?lang=en).
  % (percentage probability) | 1.1 (0.8) | 1.0 (0.5) | 1.0 (0.6)
pH (24h urine) [Mean (Full Range); unit: pH value] — Reference value: 5.50 - 7.00
  pH value | 6.13 [5.28 to 7.00] | 6.03 [4.65 to 7.14] | 6.08 [4.65 to 7.14]
pH (fasting-morning urine) [Mean (Full Range); unit: pH value] — Measure Description: Reference value 5.50 - 7.00
  pH value | 6.13 [4.97 to 7.36] | 5.87 [4.59 to 7.05] | 6.00 [4.59 to 7.36]
Potassium (24h urine) [Mean (Standard Deviation); unit: milliequivalent day-1] — Reference value: 50-100 mEq day-1
  milliequivalent day-1 | 28.60 (14.97) | 30.40 (12.98) | 29.50 (13.85)
Citrate (24h urine) [Mean (Standard Deviation); unit: mmol day-1] — Reference value: >3.3 mmol day-1
  mmol day-1 | 2.97 (1.68) | 3.50 (1.74) | 3.24 (1.71)
Citrate (fasting-morning urine) [Mean (Standard Deviation); unit: mol mol-1] — Reference value: > 0.3 mol mol-1 (Citrate/Creatinine)
  mol mol-1 | 2.77 (1.39) | 3.40 (2.39) | 3.09 (1.96)

OUTCOME MEASURES:

1. Primary Outcome: Changes in Serum Level of Carboxyterminal Cross-linked Telopeptide of Type I Collagen (CTX); Over Time, i.e. Baseline, 3 Months, 6 Months.
Description: Carboxyterminal cross-linked telopeptide of type I collagen (CTX) is a degradation product of the type I collagen; it is considered as a marker of bone resorption. The concentration of CTX (µg/L) will be measured at T0, T3, and T6 on serum samples (fasting morning samples) using commercially available reagents and following the manufacturer's protocol.
  At the end of the study, the results will be aggregated as mean ± standard of the mean, median and min-max range. Data will be statistically analyzed in order to compare the activity of Potassium citrate versus Placebo (unpaired analysis) and to evaluate the effect of Potassium Citrate and Placebo over time (paired analysis).
  Differences will be considered to be statistically significant for p-value <0.05.
Time Frame: Baseline (T0), 3 months (T3) 6 months (T6)
Population: 3/20 patients in the Treatment group did not complete the follow up (n= 1 re-evaluation of the inclusion criteria; n=1 gastritis; n=1 total hip arthroplasty).
  2/20 patients in the Placebo group did not complete the follow up (n=2 persistent constipation)
Measure: Mean (Standard Error); unit: µg/L
Arm/Group | Treatment Group, Potassium Citrate | Control Group, Placebo
Number analyzed (Participants) | 20 | 20
µg/L
  Baseline (T0) | 0.64 (0.08) | 0.64 (0.05)
  3 months (T3): number analyzed (Participants) | 18 | 20
  3 months (T3) | 0.63 (0.08) | 0.56 (0.05)
  6 months (T6): number analyzed (Participants) | 17 | 18
  6 months (T6) | 0.53 (0.08) | 0.54 (0.06)
Statistical Analysis 1: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T3 vs T0; Test type: Other; p = 0.172, t-test, 1 sided
Statistical Analysis 2: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T6 vs T0; Test type: Other; p = 0.027, t-test, 1 sided
Statistical Analysis 3: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T6 vs T3; Test type: Other; p = 0.053, t-test, 1 sided
Statistical Analysis 4: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Placebo: T3 vs T0; Test type: Other; p = 0.002, t-test, 1 sided
Statistical Analysis 5: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Placebo: T6 vs T0; Test type: Other; p = 0.006, t-test, 1 sided
Statistical Analysis 6: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Placebo: T6 vs T3; Test type: Other; p = 0.139, t-test, 1 sided
Statistical Analysis 7: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T0; Test type: Other; p = 0.967, t-test, 2 sided
Statistical Analysis 8: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T3; Test type: Other; p = 0.446, t-test, 2 sided
Statistical Analysis 9: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T6; Test type: Other; p = 0.869, t-test, 2 sided

2. Primary Outcome: Changes in Serum Levels of "Tartrate-resistant Acid Phosphatase 5b Isoenzyme" (TRAcP5b) Over Time, i.e. Baseline, 3 Months, 6 Months.
Description: Tartrate-resistant acid phosphatase 5b isoenzyme" (TRAcP5b) is a specific product of osteoclasts; it is considered as a marker of bone resorption. The concentration of TRAcP5B (U/L) will be measured at T0, T3, and T6 on serum samples (fasting morning samples) using commercially available reagents and following the manufacturer's protocol. At the end of the study, the results will be aggregated as mean ± standard of the mean, median and min-max range. Data will be statistically analyzed in order to compare the activity of Potassium Citrate versus Placebo (unpaired analysis) and to evaluate the effect of Potassium Citrate and Placebo over time (paired analysis).
  Differences will be considered to be statistically significant for p-value <0.05.
Time Frame: Baseline (T0), 3 months (T3) 6 months (T6)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: U/L
Arm/Group | Treatment Group, Potassium Citrate | Control Group, Placebo
Number analyzed (Participants) | 20 | 20
U/L
  Baseline (T0) | 2.35 (0.20) | 2.64 (0.22)
  3 months (T3): number analyzed (Participants) | 18 | 20
  3 months (T3) | 2.79 (0.27) | 2.85 (0.22)
  6 months (T6): number analyzed (Participants) | 17 | 18
  6 months (T6) | 2.69 (0.29) | 2.25 (0.14)
Statistical Analysis 1: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T3 vs T0; Test type: Other; p = 0.954, t-test, 1 sided
Statistical Analysis 2: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T6 vs T0; Test type: Other; p = 0.798, t-test, 1 sided
Statistical Analysis 3: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T6 vs T3; Test type: Other; p = 0.377, t-test, 1 sided
Statistical Analysis 4: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Placebo: T3 vs T0; Test type: Other; p = 0.886, t-test, 1 sided
Statistical Analysis 5: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Placebo: T6 vs T0; Test type: Other; p = 0.040, t-test, 1 sided
Statistical Analysis 6: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Placebo: T6 vs T3; Test type: Other; p = 0.017, t-test, 1 sided
Statistical Analysis 7: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T0; Test type: Other; p = 0.343, t-test, 2 sided
Statistical Analysis 8: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T3; Test type: Other; p = 0.859, t-test, 2 sided
Statistical Analysis 9: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T6; Test type: Other; p = 0.172, t-test, 2 sided

3. Primary Outcome: Changes in Serum Levels of "N-terminal Propeptide of Type I Procollagen" (P1NP) Over Time, i.e. Baseline, 3 Months, 6 Months.
Description: N-terminal propeptide of type I procollagen" (P1NP) is a product of the conversion of procollagen to collagen; it is considered as a marker of bone formation. The concentration of P1NP (pg/L) will be measured at T0, T3, and T6 on serum samples (fasting morning samples) using commercially available reagents and following the manufacturer's protocol. At the end of the study, the results will be aggregated as mean ± standard of the mean, median and min-max range. Data will be statistically analyzed in order to compare the activity of Potassium citrate versus Placebo (unpaired analysis) and to evaluate the effect of Potassium Citrate and Placebo over time (paired analysis).
  Differences will be considered to be statistically significant for p-value <0.05.
Time Frame: Baseline (T0), 3 months (T3) 6 months (T6)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/L
Arm/Group | Treatment Group, Potassium Citrate | Control Group, Placebo
Number analyzed (Participants) | 20 | 20
pg/L
  Baseline (T0) | 17.45 (1.48) | 18.82 (1.73)
  3 months (T3): number analyzed (Participants) | 18 | 20
  3 months (T3) | 16.24 (1.60) | 18.39 (1.75)
  6 months (T6): number analyzed (Participants) | 17 | 18
  6 months (T6) | 14.97 (1.51) | 16.77 (1.89)
Statistical Analysis 1: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T3 vs T0; Test type: Other; p = 0.213, t-test, 1 sided
Statistical Analysis 2: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T6 vs T0; Test type: Other; p = 0.191, t-test, 1 sided
Statistical Analysis 3: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T6 vs T3; Test type: Other; p = 0.234, t-test, 1 sided
Statistical Analysis 4: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Placebo: T3 vs T0; Test type: Other; p = 0.370, t-test, 1 sided
Statistical Analysis 5: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Placebo: T6 vs T0; Test type: Other; p = 0.176, t-test, 1 sided
Statistical Analysis 6: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Placebo: T6 vs T3; Test type: Other; p = 0.139, t-test, 1 sided
Statistical Analysis 7: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T0; Test type: Other; p = 0.551, t-test, 2 sided
Statistical Analysis 8: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T3; Test type: Other; p = 0.371, t-test, 2 sided
Statistical Analysis 9: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T6; Test type: Other; p = 0.466, t-test, 2 sided

4. Primary Outcome: Changes in Serum Levels of "Bone-specific Alkaline Phosphatase" (BAP) Over Time, i.e. Baseline, 3 Months, 6 Months.
Description: Bone-specific alkaline phosphatase (BAP) is a specific product of osteoblasts; it is considered as a marker of bone formation. The concentration of BAP (µg/L) will be measured at T0, T3, and T6 on serum samples (fasting morning samples) using commercially available reagents and following the manufacturer's protocol. At the end of the study, the results will be aggregated as mean ± standard of the mean, median and min-max range. Data will be statistically analyzed in order to compare the activity of Potassium citrate versus Placebo (unpaired analysis) and to evaluate the effect of Potassium Citrate and Placebo over time (paired analysis).
  Differences will be considered to be statistically significant for p-value <0.05.
Time Frame: Baseline (T0), 3 months (T3) 6 months (T6)
Population: as for outcome 1
Measure: Mean (Standard Error); unit: µg/L
Arm/Group | Treatment Group, Potassium Citrate | Control Group, Placebo
Number analyzed (Participants) | 20 | 20
µg/L
  Baseline (T0) | 21.89 (1.67) | 20.36 (1.17)
  3 months (T3): number analyzed (Participants) | 18 | 20
  3 months (T3) | 19.81 (1.67) | 18.27 (1.00)
  6 months (T6): number analyzed (Participants) | 17 | 18
  6 months (T6) | 16.83 (1.37) | 15.79 (1.09)
Statistical Analysis 1: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T3 vs T0; Test type: Other; p = 0.094, t-test, 1 sided
Statistical Analysis 2: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T6 vs T0; Test type: Other; p = 0.0004, t-test, 1 sided
Statistical Analysis 3: Comparison: Treatment Group, Potassium Citrate; Paired analysis within the group to evaluate the effect of Potassium Citrate: T6 vs T3; Test type: Other; p = 0.008, t-test, 1 sided
Statistical Analysis 4: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Placebo: T3 vs T0; Test type: Other; p = 0.002, t-test, 1 sided
Statistical Analysis 5: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Potassium Citrate: T6 vs T0; Test type: Other; p < 0.0001, t-test, 1 sided
Statistical Analysis 6: Comparison: Control Group, Placebo; Paired analysis within the group to evaluate the effect of Potassium Citrate: T6 vs T3; Test type: Other; p = 0.0007, t-test, 1 sided
Statistical Analysis 7: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T0; Test type: Other; p = 0.458, t-test, 2 sided
Statistical Analysis 8: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T3; Test type: Other; p = 0.434, t-test, 2 sided
Statistical Analysis 9: Comparison: Treatment Group, Potassium Citrate vs Control Group, Placebo; Independent comparison (unpaired analysis) between Potassium Citrate and Placebo at T6; Test type: Other; p = 0.555, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Adverse events were recorded at 3 months and 6 months
Description: Gastrointestinal disorders
Arm/Group | Treatment Group | Control Group, Placebo
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 1/20 | 2/20
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment Group (N=20) | Control Group, Placebo (N=20)
Gastritis (Gastrointestinal disorders) | 1 (1) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-03-09): https://cdn.clinicaltrials.gov/large-docs/20/NCT02731820/Prot_SAP_000.pdf